CLINICAL TRIAL: NCT05907486
Title: The Efficiency and Safety of N-acetylcysteine for Prevention of Thrombotic Events After Allogenic Hematopoietic Stem Cell Transplantation
Brief Title: The Use of N-acetylcysteine for Thrombotic Events After Allogenic Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOOCHOW-HY-2023-05-30
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Thrombotic Disorder
Keywords: Thrombotic disorder; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Thrombosis | interventions — Acetylcysteine; Busulfan; Cytarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Modified BUCY conditioning regimen: busulfan (3.2mg/kg, day-7 to day -5), cytarabine (2g/m2, day -8), cyclophosphamide (1.8g/m2, day -4 to day -3), followed by stem cells infusion; N-acetyl-cysteine (Zambon Pharma, Hainan, China) : 8g/d (>=45kg); 200mg/kg.d (<45kg), intravenously for at least 4 hours, day -9 to day +45.
  Interventions: Drug: N-acetyl-cysteine; Drug: Busulfan; Drug: Cytarabine; Drug: Cyclophosphamide
- Arm B (Active Comparator): Modified BUCY conditioning regimen: busulfan (3.2mg/kg, day-7 to day -5), cytarabine (2g/m2, day -8), cyclophosphamide (1.8g/m2, day -4 to day -3), followed by stem cells infusion.
  Interventions: Drug: Busulfan; Drug: Cytarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: N-acetyl-cysteine — 8g/d (>=45kg); 200mg/kg.d (<45kg), intravenously for at least 4 hours, day -9 to day +45
  Other Names: NAC
  Arms: Arm A
Drug: Busulfan — 3.2mg/kg, day-7 to day -5, intravenously
  Other Names: BU
Drug: Cytarabine — 2g/m2, day -8, intravenously
  Other Names: Ara-C
Drug: Cyclophosphamide — 1.8g/m2, day -4 to day -3, intravenously
  Other Names: CTX

SUMMARY:
We aim to assess the the efficiency and safety of N-acetylcysteine for prevention of thrombotic events after allogenic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
The thrombotic events are increasingly recognized complications of hematopoietic cell transplantation (HCT) associated with significant morbidity and mortality, which include transplantation-associated thrombotic microangiopathy (TA-TMA), sinusoidal obstructive syndrome (SOS), deep vein thrombosis (DVT), pulmonary thromboembolism (PTE), catheter-related thrombosis (CRT), superficial vein thrombosis (SVT), etc. There is a complex interplay on balancing the risk for thrombosis and bleeding in these patients, making treatment decisions particularly challenging. Emerging studies revealed that endothelial injury is the common underlying mechanism among different thrombotic disorders. There is increasing data that N-acetyl-cysteine (NAC) may prevent or improve endothelial dysfunction by inhibiting ROS production and preventing endothelial apoptosis. Our previous study showed low dose NAC could decrease the incidence of TA-TMA. In this study, we aim to assess the the efficiency and safety of N-acetylcysteine for prevention of thrombotic events after allogenic hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16-70 years old
2. Diagnosed as myeloid malignancies, and about to undergo allo-HSCT;
3. ECOG: 0-2;
4. Expected survival longer than 1 month

Exclusion Criteria:

1. Allergic to any components of NAC;
2. Severe dysfunction of heart, liver, lung and kidney;
3. Relapse before HSCT;
4. A history of bronchial asthma, bronchospasm or moderate / severe gastrohelcosis.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of thrombotic disorders | 1 year
  The incidence of thrombotic disorders (TA-TMA, SOS, DVT, PTE, CRT, SVT) after allogenic hematopoietic stem cell transplantation
Overall survival | 1 year
  The rate of overall survival after allogenic hematopoietic stem cell transplantation

SECONDARY OUTCOMES:
The incidence of relapse | 1 year
  The incidence of relapse after allogenic hematopoietic stem cell transplantation
The incidence of GVHD | 1 year
  The incidence of GVHD after allogenic hematopoietic stem cell transplantation
The incidence of hematopoietic reconstitution | 1 year
  The incidence of hematopoietic reconstitution after allogenic hematopoietic stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, Professor, Study Chair — The First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labrador J, Lopez-Anglada L, Perez-Lopez E, Lozano FS, Lopez-Corral L, Sanchez-Guijo FM, Vazquez L, Perez Rivera JA, Martin-Herrero F, Sanchez-Barba M, Guerrero C, del Canizo MC, Caballero MD, San Miguel JF, Alberca I, Gonzalez-Porras JR. Analysis of incidence, risk factors and clinical outcome of thromboembolic and bleeding events in 431 allogeneic hematopoietic stem cell transplantation recipients. Haematologica. 2013 Mar;98(3):437-43. doi: 10.3324/haematol.2012.069559. Epub 2012 Aug 16. PMID 22899581
- [Background] Laskin BL, Goebel J, Davies SM, Jodele S. Small vessels, big trouble in the kidneys and beyond: hematopoietic stem cell transplantation-associated thrombotic microangiopathy. Blood. 2011 Aug 11;118(6):1452-62. doi: 10.1182/blood-2011-02-321315. Epub 2011 May 19. PMID 21596850
- [Background] George JN, Li X, McMinn JR, Terrell DR, Vesely SK, Selby GB. Thrombotic thrombocytopenic purpura-hemolytic uremic syndrome following allogeneic HPC transplantation: a diagnostic dilemma. Transfusion. 2004 Feb;44(2):294-304. doi: 10.1111/j.1537-2995.2004.00700.x. PMID 14962323
- [Background] Coppell JA, Richardson PG, Soiffer R, Martin PL, Kernan NA, Chen A, Guinan E, Vogelsang G, Krishnan A, Giralt S, Revta C, Carreau NA, Iacobelli M, Carreras E, Ruutu T, Barbui T, Antin JH, Niederwieser D. Hepatic veno-occlusive disease following stem cell transplantation: incidence, clinical course, and outcome. Biol Blood Marrow Transplant. 2010 Feb;16(2):157-68. doi: 10.1016/j.bbmt.2009.08.024. Epub 2009 Sep 18. PMID 19766729
- [Background] Tsirigotis PD, Resnick IB, Avni B, Grisariu S, Stepensky P, Or R, Shapira MY. Incidence and risk factors for moderate-to-severe veno-occlusive disease of the liver after allogeneic stem cell transplantation using a reduced intensity conditioning regimen. Bone Marrow Transplant. 2014 Nov;49(11):1389-92. doi: 10.1038/bmt.2014.168. Epub 2014 Jul 28. PMID 25068424
- [Background] Carreras E, Diaz-Beya M, Rosinol L, Martinez C, Fernandez-Aviles F, Rovira M. The incidence of veno-occlusive disease following allogeneic hematopoietic stem cell transplantation has diminished and the outcome improved over the last decade. Biol Blood Marrow Transplant. 2011 Nov;17(11):1713-20. doi: 10.1016/j.bbmt.2011.06.006. Epub 2011 Jun 25. PMID 21708110
- [Background] Jodele S, Laskin BL, Dandoy CE, Myers KC, El-Bietar J, Davies SM, Goebel J, Dixon BP. A new paradigm: Diagnosis and management of HSCT-associated thrombotic microangiopathy as multi-system endothelial injury. Blood Rev. 2015 May;29(3):191-204. doi: 10.1016/j.blre.2014.11.001. Epub 2014 Nov 28. PMID 25483393
- [Background] Ho VT, Cutler C, Carter S, Martin P, Adams R, Horowitz M, Ferrara J, Soiffer R, Giralt S. Blood and marrow transplant clinical trials network toxicity committee consensus summary: thrombotic microangiopathy after hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2005 Aug;11(8):571-5. doi: 10.1016/j.bbmt.2005.06.001. PMID 16041306
- [Background] Sartain S, Shubert S, Wu MF, Srivaths P, Teruya J, Krance R, Martinez C. Therapeutic Plasma Exchange does not Improve Renal Function in Hematopoietic Stem Cell Transplantation-Associated Thrombotic Microangiopathy: An Institutional Experience. Biol Blood Marrow Transplant. 2019 Jan;25(1):157-162. doi: 10.1016/j.bbmt.2018.08.016. Epub 2018 Aug 23. PMID 30144562